CLINICAL TRIAL: NCT04643002
Title: Phase 1-2 UMBRELLA Trial Evaluating Isatuximab With or Without Dexamethasone in Combination With Novel Agents Compared to Isatuximab With Pomalidomide and Dexamethasone in Relapsed or Refractory Multiple Myeloma (RRMM) - Master Protocol
Brief Title: Isatuximab in Combination With Novel Agents in RRMM - Master Protocol
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16482; U1111-1244-2598 (Registry Identifier: ICTRP); 2024-514988-25 (Registry Identifier: CTIS); 2020-003024-16 (EudraCT Number)
Record Dates: First submitted 2020-10-20; First posted 2020-11-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Plasma Cell Myeloma Refractory
Keywords: anti-CD38 monoclonal antibody; master protocol; combination therapy; CD38 resistance; interleukin 2; ROCK2 inhibitor; anti-CD47 agent
MeSH Terms: interventions — isatuximab; Dexamethasone; pomalidomide; belantamab mafodotin; belumosudil; ALX148

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Control Arm: isatuximab + pomalidomide + dexamethasone (Substudy 01) (Active Comparator): * Isatuximab, intravenous (IV) doseweekly (QW) × 4 weeks (Cycle 1), followed by every two weeks (Q2W) (subsequent cycles).
  * Pomalidomide dose by mouth daily Day 1 to Day 21.
  * Dexamethasone dose by mouth QW.
  Interventions: Drug: Isatuximab; Drug: Dexamethasone; Drug: Pomalidomide
- isatuximab + SAR439459 + dexamethasone (Substudy 02) (Experimental): SAR439459 in combination with isatuximab and dexamethasone
  Part 1:
  2 dose levels (DLs) of IV SAR439459:
  * DL1 SAR439459 dose Q2W.
  * DL2 SAR439459 dose Q2W.
  * Isatuximab dose IV QW × 5 weeks (Cycle 1), followed by Q2W administrations (subsequent cycles).
  * Dexamethasone fixed dose and schedule: QW by mouth In Cycle 1, the first administration of SAR439459 (Day 1) will precede isatuximab by 1 week (first dose of isatuximab will be at Cycle 1 Day 8).
  Part 2:
  * SAR439459 IV dose Q2W.
  * Isatuximab IV dose QW × 5 weeks (Cycle 1), followed by Q2W administrations (subsequent cycles).
  * Dexamethasone fixed dose and schedule: QW by mouth. In Cycle 1, the first administration of SAR439459 (Day 1) will precede isatuximab by 1 week (first dose of isatuximab will be at Cycle 1 Day 8).
  Interventions: Drug: Isatuximab; Drug: Dexamethasone; Drug: SAR439459
- isatuximab + dexamethasone + belantamab mafodotin (Substudy 03) (Experimental): Belantamab mafodotin in combination with isatuximab and dexamethasone
  Part 1:
  1 DL of IV belantamab mafodotin in Part 1 and de-escalation dose DL-1:
  * DL1 belantamab mafodotin IV dose QW4 or de-escalation dose DL-1 QW8
  * Isatuximab dose, IV QW × 4 weeks (Cycle 1), followed by Q2W (subsequent cycles).
  * Dexamethasone fixed dose and schedule: QW by mouth.
  Part 2:
  * Isatuximab IV dose QW × 4 weeks (Cycle 1), followed by Q2W (subsequent cycles).
  * Belantamab mafodotin IV dose Q4W or Q8W
  * Dexamethasone fixed dose and schedule: QW by mouth.
  Interventions: Drug: Isatuximab; Drug: Dexamethasone; Drug: Belantamab mafodotin
- Isatuximab + pegenzileukin (Substudy 04) (Experimental): Pegenzileukin in combination with isatuximab
  Part 1- dose escalation:
  * Up to 3 DLs of IV pegenzileukin are planned to be evaluated:
    * DL1 will explore pegenzileukin at Q2W.
    * DL2 will explore pegenzileukin at Q2W.
    * DL3 will explore pegenzileukin at Q2W.
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles).
  Part 1 - dose optimization:
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles).
  * Pegenzileukin at potential doses (DL A and DL B) Q2W.
  Part 2 (dose expansion):
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles).
  * Pegenzileukin IV dose Q2W.
  Interventions: Drug: Isatuximab; Drug: Pegenzileukin
- Experimental: Isatuximab + Dexamethasone + Belumosudil (Substudy 05) (Experimental): Isatuximab in combination with belumosudil and dexamethasone Part 1- dose escalation: During the first cycle, belumosudil will be evaluated in monotherapy during 2 to 4 weeks, then isatuximab and dexamethasone will be added, and continued for the subsequent cycles.
  * Belumosudil by mouth at Dose Level (DL) 1, DL2, DL3, and DL4
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles)
  * Dexamethasone fixed dose and schedule: QW by mouth
  Part 1- dose optimization:
  * Belumosudil at potential doses (DL A and DL B), daily by mouth
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles)
  * Dexamethasone fixed dose and schedule: QW by mouth
  Part 2- dose expansion:
  * Belumosudil dose daily, by mouth
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles)
  * Dexamethasone fixed dose and schedule: QW by mouth
  Interventions: Drug: Isatuximab; Drug: Dexamethasone; Drug: Belumosudil
- Isatuximab + evorpacept + dexamethasone (Substudy 06) (Experimental): Isatuximab in combination with evorpacept and dexamethasone
  Part 1- dose escalation:
  * Evorpacept IV dose Q2W
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles)
  * Dexamethasone fixed dose and schedule: QW by mouth Part 1- dose optimization
  * Evorpacept IV at potential doses (DL A and DL B), Q2W
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles)
  * Dexamethasone fixed dose and schedule: QW by mouth
  Part 2- dose expansion:
  * Evorpacept IV dose Q2W
  * Isatuximab IV dose QW × 4 weeks, followed by Q2W (subsequent cycles)
  * Dexamethasone fixed dose and schedule: QW by mouth
  Interventions: Drug: Isatuximab; Drug: Dexamethasone; Drug: Evorpacept

INTERVENTIONS:
Drug: Isatuximab — Pharmaceutical form: Concentrated solution for intravenous infusion; Route of administration: Intravenous infusion
  Other Names: SAR650984; Sarclisa®
Drug: Dexamethasone — Pharmaceutical form: Tablet; Route of administration: Oral
  Arms: Control Arm: isatuximab + pomalidomide + dexamethasone (Substudy 01); Experimental: Isatuximab + Dexamethasone + Belumosudil (Substudy 05); Isatuximab + evorpacept + dexamethasone (Substudy 06); isatuximab + SAR439459 + dexamethasone (Substudy 02); isatuximab + dexamethasone + belantamab mafodotin (Substudy 03)
Drug: Pomalidomide — Pharmaceutical form: Capsule; Route of administration: Oral
  Other Names: Pomalyst®
  Arms: Control Arm: isatuximab + pomalidomide + dexamethasone (Substudy 01)
Drug: Belantamab mafodotin — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Other Names: BLENREP®
  Arms: isatuximab + dexamethasone + belantamab mafodotin (Substudy 03)
Drug: Pegenzileukin — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Other Names: SAR444245
  Arms: Isatuximab + pegenzileukin (Substudy 04)
Drug: SAR439459 — Pharmaceutical form: Solution for injection; Route of administration: Intravenous
  Arms: isatuximab + SAR439459 + dexamethasone (Substudy 02)
Drug: Belumosudil — Pharmaceutical form: tablet; route of administration: oral
  Other Names: SAR445761,; Rezurock
  Arms: Experimental: Isatuximab + Dexamethasone + Belumosudil (Substudy 05)
Drug: Evorpacept — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Other Names: ALX148
  Arms: Isatuximab + evorpacept + dexamethasone (Substudy 06)

SUMMARY:
The purpose of this umbrella study is to evaluate isatuximab when combined with novel agents with or without dexamethasone in participants with relapsed or refractory myeloma. Substudy 01 is the control Substudy. Substudies 02, 03, and 06 are controlled experimental substudies. Substudies 04 and 05 are independent experimental substudies.

DETAILED DESCRIPTION:
Participants will continue study treatment until disease progression, death, unacceptable toxicity, participant request to stop treatment, Investigator decision, or study termination by the Sponsor i.e., up to Aapproximately 28 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive or older.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Participants with relapsed or refractory MM who have received at least 2 prior lines of therapy for MM, including PIs and IMiDs (eg, Induction regimen with autologous stem cell transplant followed by maintenance is considered one line).
* RRMM with measurable disease:

  * Serum M protein ≥0.5 g/dL measured using serum protein immunoelectrophoresis and/or
  * Urine M protein ≥200 mg/24 hours measured using urine protein immunoelectrophoresis and/or
  * Serum free light chain (sFLC) MM without measurable M protein in serum or urine per previous criteria (serum Ig free light chain ≥10 mg/dL and abnormal serum Ig kappa lambda free light chain ratio <0.26 or >1.65).
* Men or woman or childbearing potential should agree to use contraception.
* Substudy 01, 06: Anti-CD38 therapy naïve or prior exposure to such drugs with a wash out of at least 12 months after the last dose. "Exposure" is defined as at least 2 cycles of therapy.
* Substudies 02, 03: Anti-CD38 therapy naïve or prior exposure to such drugs without being refractory but with a wash out of at least 6 months after the last dose. "Refractory" is defined as progressing within 60 days of last dose of anti-CD38 targeting therapy.
* Substudy 04: Anti-CD38 and anti-B cell maturation antigen (BCMA) therapy (if available) prior exposed participants with RRMM. For anti-CD38, "Exposure" is defined as at least 2 cycles of therapy. For anti-BCMA therapy if available, exposure is defined by at least 2 cycles of therapy.
* Substudy 05: Participants with RRMM with at least 2 cycles of prior exposure to anti-CD38 therapy. For participants to whom BCMA targeted therapy is available (ie, approved in their region and can be reimbursed), at least 2 cycles of prior exposure to a BCMA targeted agent is mandatory.

Exclusion Criteria:

* Primary systemic amyloid light chain amyloidosis, plasma cell leukemia, monoclonal gammopathy of undetermined significance, or smoldering myeloma.
* Uncontrolled infection within 14 days prior to first study intervention administration.
* Clinically significant cardiac (including valvular) or vascular disease within 3 months prior to first study intervention administration., eg, myocardial infarction, unstable angina, coronary (eg, coronary artery bypass graft, percutaneous coronary intervention) or peripheral artery revascularization, left ventricular ejection fraction <40%, heart failure New York Heart Association Classes III and IV, stroke, transient ischemic attack, pulmonary embolism, other thromboembolic event, or cardiac arrhythmia (Grade 3 or higher by NCI CTCAE Version 5.0).
* Known acquired immunodeficiency syndrome-related illness or known human immunodeficiency virus (HIV) disease requiring antiviral treatment or active hepatitis A.
* Uncontrolled or active hepatitis B virus (HBV) infection.
* Active hepatitis C virus (HCV) infection.
* Any of the following within 3 months prior to first study intervention administration: treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease.
* Second malignancy other than basal cell or squamous cell carcinoma of the skin or in situ carcinoma, unless they are successfully treated with curative intent for more than 3 years before first study intervention administration.
* Any anti-MM drug treatment within 14 days before first study intervention administration, including dexamethasone.
* Participants with a contraindication to treatment.
* Vaccination with a live vaccine 4 weeks before the start of the study.
* Seasonal flu and COVID-19 vaccines that do not contain live virus are permitted.
* Hemoglobin <8 g/dL.
* Platelets <50 × 10^9/L.
* Absolute neutrophil count <1.0 × 10^9/L.
* Creatinine clearance <30 mL/min/1.73m2.
* Total bilirubin >1.5 × ULN, except for known Gilbert syndrome in which direct bilirubin should be ≤2.5 × ULN.
* Aspartate aminotransferase and/or alanine aminotransferase >3 × ULN.
* Patients with grade 3 or 4 hypercalcemia.

Substudy 01:

-Malabsorption syndrome or any condition that can significantly impact the absorption of pomalidomide.

Substudy 02:

* History of resected/ablated basal or squamous cell carcinoma (SCC) of the skin or carcinoma in situ of the cervix, or other local tumors, even if considered cured by local treatment.
* Therapeutic doses of anticoagulants or antiplatelet agents within 7 days prior to the first dose of SAR439459.
* Prothrombin time or INR >1.5 × upper limit of normal (ULN).

Substudy 03:

* Current corneal epithelial disease except mild punctate keratopathy.
* Patients who have received prior therapy with belantamab mafodotin.

Substudy 04:

* Central nervous system or leptomeningeal disease.
* Medical history of seizure.
* Participants currently receiving hepatically metabolized narrow therapeutic index drugs (eg, digoxin, warfarin) if cannot be closely monitored.
* Active, known, or suspected autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs), except controlled by replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc). The following are not exclusionary: vitiligo, childhood asthma that has resolved, psoriasis that does not require systemic treatment.
* Prior allogeneic hematopoietic stem cell transplant (allo-HSCT).

Substudy 05:

- Participant unable to swallow tablets.

Substudy 06:

* History of active autoimmune disorders.
* History of autoimmune hemolytic anemia or autoimmune. thrombocytopenia.
* Active graft versus host disease (GVHD) or ongoing immunosuppression for GVHD.
* Prior allogenic hematopoietic stem cell transplant (allo-HSCT).
* Patient with chronic active EBV infection.
* Patients with known history of HLH.
* Hemoglobin < 9 g/dL.
* Prior therapy with any anti-CD47 or anti signal regulatory protein alpha agent.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2027-09-13 (Estimated); Study Completion 2028-04-20 (Estimated)

PRIMARY OUTCOMES:
Part 1 (dose finding, experimental substudies): Determination of recommended dose of novel agents in combination with isatuximab | Through the end of cycle 1 (approximately 6 weeks)
  Determination or confirmation of the dose will be based on: safety and tolerability in terms of TEAEs/SAEs, dose-limiting toxicity occurrence, and laboratory parameters available information on PK (if appropriate) and biomarkers.
Part 2 (expansion, controlled experimental substudies): VGPR Rate (Rate of Very Good Partial Response Rate or Better) | Up to approximately 28 months after the First patient in or scheduled assessment
  VGPR or better rate is defined as the percentage of participants with a VGPR or better as defined by the 2016 IMWG response criteria, assessed by Investigator based on central laboratory values and local imaging.
Part 2 (expansion, independent experimental substudies): Overall Response Rate (ORR) in independent experimental substudies | Up to approximately 28 months after the First patient in or scheduled assessment
  ORR, defined as the proportion of participants with stringent complete response (sCR), complete response (CR), VGPR, or partial response (PR), according to the 2016 IMWG criteria assessed by Investigator based on central laboratory values and local imaging.

SECONDARY OUTCOMES:
Part 1 (dose finding, experimental substudies): ORR | Up to approximately 28 months after the First patient in or scheduled assessment
  ORR, defined as the proportion of participants with stringent complete response (sCR), complete response (CR), VGPR, or partial response (PR), according to the 2016 IMWG criteria assessed by Investigator based on central laboratory values and local imaging.
Part 2 (expansion, controlled experimental substudies): ORR | Up to approximately 28 months after the First patient in or scheduled assessment
  ORR, defined as the proportion of participants with stringent complete response (sCR), complete response (CR), VGPR, or partial response (PR), according to the 2016 IMWG criteria assessed by Investigator based on central laboratory values and local imaging.
Part 1 (dose finding, experimental substudies): VGPR or better | Up to approximately 28 months after the First patient in or scheduled assessment
  VGPR or better rate is defined as the percentage of participants with a VGPR or better as defined by the 2016 IMWG response criteria, assessed by Investigator based on central laboratory values and local imaging.
Part 2 (expansion, independent experimental substudies): VGPR or better | Up to approximately 28 months after the First patient in or scheduled assessment
  VGPR or better rate is defined as the percentage of participants with a VGPR or better as defined by the 2016 IMWG response criteria, assessed by Investigator based on central laboratory values and local imaging.
Clinical benefit rate (CBR) in each treatment arm | Up to approximately 28 months after the First patient in or scheduled assessment
  CBR, defined as the proportion of participants with sCR, CR, VGPR, PR, or minimal response, according to the 2016 IMWG criteria assessed by Investigator based on central laboratory values and local imaging.
Duration of Response (DOR) in each treatment arm | Up to approximately 28 months after the First patient in or scheduled assessment
  DOR, defined as the time from the date of the first response that is subsequently confirmed for patients achieving PR or better to the date of first documented PD or death, whichever happens first.
Time to First Response (TT1R) in each treatment arm | Up to approximately 28 months after the First patient in or scheduled assessment
  TT1R, defined as the time from the date of first treatment to the date of first response (PR or better) that is subsequently confirmed.
Time to Best Response (TTBR) in each treatment arm | Up to approximately 28 months after the First patient in or scheduled assessment
  TTBR, defined as the time from the date of first treatment to the date of first occurrence of best overall response (PR or better) that is subsequently confirmed.
Number of participants with treatment emergent adverse events and serious adverse events in each treatment arm | Up to approximately 28 months after the First patient in or scheduled assessment
  Safety and tolerability assessed in terms of adverse events/SAEs, including second primary malignancies, laboratory parameters, vital signs, and findings from physical examination.
Progression-free survival (PFS) in each treatment arm | Up to approximately 28 months after the First patient in or scheduled assessment
  PFS is defined as the time from the date of first treatment to disease progression based on the Investigator assessment according to 2016 IMWG criteria or death from any cause, whichever happens first.
Overall Survival (OS) in each treatment arm | Up to approximately 28 months after the First patient in or scheduled assessment
  OS is defined as the time from the date of first treatment to death from any cause.
Immunogenicity of isatuximab and novel agents | Multiple timepoints up to approximately 28 months after the First patient in or scheduled assessment
  Incidence of anti-drug antibodies (ADAs) for novel agents (experimental arms) and isatuximab.
Concentration of novel agents (experimental arms) and isatuximab (Ctrough) | Multiple timepoints during Cycle 1. The cycle is 28 days.
Disease-specific HRQL will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) core quality of life questionnaire (QLQ-C30) | On Day1 Cycle 1, then every 2 cycles for the first year; then every 3 cycles thereafter, at end of treatment and at first follow-up visit. The cycle is 28 days.
  The EORTC QLQ-C30 will be used to assess cancer-specific HRQL, disease and treatment-related symptoms and impact of symptoms. This endpoint will be assessed for Part 1 (dose optimization, independent and controlled experimental substudies) and Part 2 (expansion, independent and controlled experimental substudies).
Disease- and treatment-related quality of life will be assessed using the EORTC multiple myeloma module (QLQ-MY20) questionnaire | On Day1 Cycle 1, then every 2 cycles for the first year; then every 3 cycles thereafter, at end of treatment and at first follow-up visit. The cycle is 28 days.
  The EORTC QLQ-MY20 will be used to measure myeloma-specific HRQL, disease and treatment-related symptoms and impact of symptoms. This endpoint will be assessed for Part 1 (dose optimization, independent and controlled experimental substudies) and Part 2 (expansion, independent and controlled experimental substudies).
Global impact of side effects will be assessed using the Functional Assessment of Cancer Therapy (FACT-G) (GP5) | On Day1 Cycle 1, then every 2 cycles for the first year; then every 3 cycles thereafter, at end of treatment and at first follow-up visit. The cycle is 28 days.
  A single item from the FACT-G GP5 will be used to assess the global impact of side effects. This endpoint will be assessed for Part 1 (dose optimization, independent and controlled experimental substudies) and Part 2 (expansion, independent and controlled experimental substudies).
Estimate/Confirm established clinically meaningful change scores for clinical outcome assessments (COAs)/domain scores using the Patient Global Impression of Severity (PGIS) and Patient Global Impression of Change (PGIC) scales | On Day1 Cycle 1, then every 2 cycles for the first year; then every 3 cycles thereafter, at end of treatment and at first follow-up visit. The cycle is 28 days.
  Patient Global Impression of Severity (PGIS) and Patient Global Impression of Change (PGIC) scales will be utilized as anchors to estimate/confirm established clinically meaningful change scores for clinical outcome assessments (COAs)/domain scores. This endpoint will be assessed for Part 1 (dose optimization, independent and controlled experimental substudies) and Part 2 (expansion, independent and controlled experimental substudies).
The intensity of skeletal-related events (SRE)- related bone pain will be assessed using the skeletal-related bone pain numeric rating scale (SRE-BP-NRS) for control and experimental arms -Substudy 02 | On Day1 Cycle 1, then every 2 cycles for the first year; then every 3 cycles thereafter, at end of treatment and at first follow-up visit. The cycle is 28 days.
  The SRE-BP-NRS) will be used to assess the intensity of SRE-related bone pain (on average and at its worst) for control arm only
SRE Incidence for control and experimental arms- Substudy 02 | Continuous throughout study assessment (up to approximately 28 months)
  SRE incidence, defined as the proportion of participants who experienced pathological fracture, radiation to bone, spinal cord compression, or surgery to bone as a first bone event.
Time to First Occurrence of SRE Assessment for control and experimental arms (Substudy 02) | Continuous throughout study assessment (up to approximately 28 months)
  Time to first occurrence of SRE is defined as time from the date of randomization to the occurrence of first SRE.
Assessment of Health care resource utilization related with SREs for control and experimental arms -Substudy 02 | On Day1 Cycle 1, then every 2 cycles for the first year; then every 3 cycles thereafter, at End of treatment and at first follow-up visit. The cycle is 28 days.
  The Health Care Resource Use-SREs questionnaire (HCRU-SREs) will be used to assess the use of health care resources associated with these events.
To assess patient-reported visual functioning for experimental arm only -Substudy 03 | On Day1 Cycle 1, End of treatment and at first follow-up visit. The cycle is 28 days.
  An NEI VFQ-25 will be used to assess patient-reported visual functioning.
Maximum concentration observed after the first infusion (Cmax) for Belumosudil - Substudy 05 | Multiple timepoints during Cycle 1. The cycle is 28 days.
Time to reach Cmax (tmax) for Belumosudil - Substudy 05 | Multiple timepoints during Cycle 1. The cycle is 28 days.
Area under the concentration versus time curve calculated using the trapezoidal method from 0 to 8h (AUC0-8h) for Belumosudil - Substudy 05 | Multiple timepoints during Cycle 1. The cycle is 28 days.
Maximum concentration observed after the first infusion (Cmax) for Evorpacept - Substudy 06 | Multiple timepoints during Cycle 1. The cycle is 28 days.
Time to reach Cmax (tmax) for Evorpacept - Substudy 06 | Multiple timepoints during Cycle 1. The cycle is 28 days.
Area under the concentration versus time curve calculated using the trapezoidal method over the dosing interval for evorpacept (AUC0-t)- Substudy 06 | Multiple timepoints during Cycle 1. The cycle is 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (27):
- United States (4):
  - Winship Cancer Institute, Emory University- Site Number : 8400010, Atlanta, Georgia
  - University of Illinois-Chicago - College of Medicine- Site Number : 8400007, Chicago, Illinois
  - University of Michigan Health System - Ann Arbor- Site Number : 8400004, Ann Arbor, Michigan
  - Roswell Park Cancer Institute- Site Number : 8400008, Buffalo, New York
- Australia (3):
  - Investigational Site Number : 0360006, Wollongong, New South Wales
  - Investigational Site Number : 0360002, Melbourne, Victoria
  - Investigational Site Number : 0360001, Richmond, Victoria
- France (4):
  - Investigational Site Number : 2500002, Lille
  - Investigational Site Number : 2500001, Nantes
  - Investigational Site Number : 2500004, Paris
  - Investigational Site Number : 2500003, Paris
- Germany (2):
  - Investigational Site Number : 2760006, Frankfurt
  - Investigational Site Number : 2760008, Lübeck
- Greece (2):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000001, Athens
- Israel (3):
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760003, Ramat Gan
  - Investigational Site Number : 3760001, Tel Aviv
- Investigational Site Number : 3800001, Meldola, Reggio Emilia, Italy
- Investigational Site Number : 5780001, Oslo, Norway
- Portugal (2):
  - Investigational Site Number : 6200001, Coimbra
  - Investigational Site Number : 6200002, Porto
- Puerto Rico Medical Research Center- Site Number : 8400005, HATO REY, Puerto Rico, Puerto Rico
- South Korea (4):
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org